CLINICAL TRIAL: NCT01094392
Title: Influence on Hemostasis During Prolonged Asparaginase Treatment in Childhood and Adolescent ALL
Brief Title: Hemostasis During Asparaginase Treatment in Acute Lymphoblastic Leukemia(ALL)
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Birgitte Klug Albertsen, MD, PhD, Aarhus University Hospital
Other Study IDs: Hemostasis-NOPHO
Record Dates: First submitted 2010-03-17; First posted 2010-03-29 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2016-03

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL; PEG-asparaginase; prolonged treatment; Thrombosis; Central venous line; Echocardiography
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- treatment every 6th week during 6 months
- treatment every 2nd week during 6 months

SUMMARY:
Asparaginase is an important drug in the treatment of childhood leukemia. One of the rare but severe side effects to the treatment is thrombosis in or outside the central nervous system.

The aim of this study is to investigate and describe the influence on the coagulation parameters during prolonged treatment with asparaginase.

Hopefully this knowledge will help to foresee the risk of thrombosis and thus making it possible to prevent these.

ELIGIBILITY:
Inclusion Criteria:

* Childhood ALL, eligible to receive standard risk or intermediate risk therapy as described in the protocol, written informed consent has been obtained

Exclusion Criteria:

* No allergic reactions to PEG-asparaginase

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young adults (age 1-17.9 years) newly diagnosed with ALL in the Nordic Countries and treated according to the Nordic ALL-protocol NOPHO ALL-2008.
  Written informed consent has been obtained
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2010-03; Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Description of the coagulation parameters | December 2016
  The study is a prospective and descriptive study. Levels of coagulation parameters will be analyzed using Two Sample T-Test and the levels of asparaginase in serum will be analyzed by Chi2 test.

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte K Albertsen, Ph.D. M.D., Principal Investigator — Department of Pediatrics, Skejby Hospital, Aarhus, Denmark
Locations (4):
- Denmark (4):
  - Aalborg Hospital, Aalborg
  - Department of Pediatrics, Skejby Hospital, Aarhus
  - Department of Pediatrics, Rigshospitalet, Copenhagen
  - University Hospital in Odense, Odense